CLINICAL TRIAL: NCT02323373
Title: Topical Versus Intravenous Tranexamic Acid in Total Knee Arthroplasty: a Randomized Clinical Trial With 90 Patients
Brief Title: Topical Versus Intravenous Tranexamic Acid in Total Knee Arthroplasty
Acronym: TRANEXTKA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Ari Zekcer, MD, PhD, Irmandade da Santa Casa de Misericordia de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ISCMSP
Record Dates: First submitted 2014-12-10; First posted 2014-12-23 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Arthrosis
Keywords: Arthroplasty, Replacement, Knee; Tranexamic Acid; Drug Administration Routes
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical group (Experimental): Intervention: Tranexamic Acid - topical. Topical administration of a solution of 1.5 g of tranexamic acid (50 mg/ml, Transamin, Zydus Nikkho) diluted in 50 ml of saline (at 0.9%), sprayed over the operated area, covering it for 5 minutes, before the tourniquet release.
  Interventions: Drug: Tranexamic Acid - topical
- Intravenous group (Active Comparator): Intervention: Tranexamic Acid - intravenous Intravenous injection of 20 mg/kg of tranexamic acid, diluted in 100 ml of saline at 0.9%, administered with anesthesia in 10 minutes.
  Interventions: Drug: Tranexamic Acid - intravenous
- Placebo (Placebo Comparator): Intervention: intravenous injection of 100 ml of saline solution also administered with anesthesia in 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid - topical — Tranexamic acid is an antifibrinolytic agent that decreases perioperative blood loss, because it inhibits fibrinolysis by competing with lysine molecule in coupling sites in fibrinogen. In this study arm, the drug is administered topically on the wound.
  Other Names: trans-4-(aminomethyl)cyclohexanecarboxylic acid
  Arms: Topical group
Drug: Placebo — 100 ml of saline solution administered with anesthesia during 10 minutes
  Other Names: Saline solution
  Arms: Placebo
Drug: Tranexamic Acid - intravenous — Tranexamic acid is an antifibrinolytic agent that decreases perioperative blood loss, because it inhibits fibrinolysis by competing with lysine molecule in coupling sites in fibrinogen. In this arm, the drug is administered intravenously.
  Other Names: trans-4-(aminomethyl)cyclohexanecarboxylic acid
  Arms: Intravenous group

SUMMARY:
This clinical trial investigated two different routes of administration of tranexamic acid in total knee arthroplasty: topical compared to intravenous.

DETAILED DESCRIPTION:
Intravenous administration of tranexamic acid (TA) is common in orthopedic surgery. The ideal dose and administration route of the drug in total knee arthroplasty (TKA) is under investigation.

The objective of this randomized clinical trial was to verify differences between topical and intravenous administration of TA in TKA regarding blood loss and coagulation variables.

Patients undergoing TKA were randomized to receive TA intravenously (20 mg in 100 ml of saline), topically (1.5 g in 50 ml of saline, sprayed over the operated site, before closure) or intravenous saline (100 ml). Suction drains were maintained for 48 hours, in order to measure blood loss. Data analysis is being undertaken now, in order to compare the two routes of administration of the drug.

ELIGIBILITY:
Inclusion Criteria: Patients in need of unilateral total knee arthroplasty (TKA) due to arthrosis, Albach grades III and IV were eligible

Exclusion Criteria:

* history or identified risk for deep vein thrombosis or pulmonary embolism
* history of coagulation or cardiovascular disorders
* vascular diseases
* pregnancy
* current use of anticoagulation drugs
* previous orthopedic surgery in the legs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Blood loss | up to 48 hours from the end of surgery, with drained volume registered every 6 hours.
  Volume of blood loss in the suction drain device after TKA surgery

SECONDARY OUTCOMES:
Thrombosis | up to 15 days after surgery
  Patients with events of thrombosis after TKA
Need for transfusion | during or after surgery, during hospital stay (hospital discharge took place in four days, in average)
  Number (or percentage) of patients requiring transfusion in TKA surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zekcer Ari, MD, PhD, Principal Investigator — Santa Casa de São Paulo